CLINICAL TRIAL: NCT04927611
Title: Single-cell Sequencing and Establishment of Cell Lines, Organoids, and Transplanted Tumor Models in Neuroendocrine Neoplasm
Brief Title: Single-cell Sequencing and Establishment of Models in Neuroendocrine Neoplasm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: D1 Medical Technology (Shanghai) Co., Ltd, China (Industry)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Shanghai Pancreatic Cancer Institute, Fudan University
Other Study IDs: CSPAC-NEN-1
Record Dates: First submitted 2021-06-02; First posted 2021-06-16 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Neuroendocrine Neoplasm
Keywords: Neuroendocrine Neoplasm; Single Cell Sequencing Technology; Primary Cell Culture; Organoid; Patient-derived Tumor Xenograft
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Biopsy; Laparoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastroenteropancreatic neuroendocrine neoplasms: Collect biopsy/surgical fresh tissue of gastroenteropancreatic neuroendocrine neoplasms.
  Interventions: Procedure: Biopsy, open or laparoscopic surgery
- Pancreatic ductal adenocarcinoma: Collect biopsy/surgical fresh tissue of pancreatic ductal adenocarcinoma.
  Interventions: Procedure: Biopsy, open or laparoscopic surgery

INTERVENTIONS:
Procedure: Biopsy, open or laparoscopic surgery — Collect NEN and PDAC biopsy or surgical fresh tissue to conduct single cell sequencing or model construction.

SUMMARY:
The aim of this study is to use single-cell sequencing technology to explore neuroendocrine neoplasm (NEN) molecular biological characteristics, tumor heterogeneity and cell subtypes. Besides. NEN models are constructed for basic research, including primary cell lines, organoids, and animal models.

DETAILED DESCRIPTION:
Neuroendocrine neoplasm (NEN) generally refers to all tumors that originate from peptidergic neurons and neuroendocrine cells. It is a relatively rare tumor, ranging from indolent, slow-growing low-grade malignant tumors to obvious distant metastases. A series of malignant tumors. The most common place for neuroendocrine tumors is in the digestive system, and about two-thirds of neuroendocrine tumors occur in the gastrointestinal pancreas. However, with the change of people's living habits and the improvement of physical examination awareness, the incidence of neuroendocrine tumors increased from 1.09/100,000 in 1973 to 6.98/100,000 in 2012. The incidence has increased by 6 times compared with other tumors. , NENs increase more rapidly. The incidence of people over 65 years of age has increased by 8 times, and the incidence of people younger than 50 years of age has also increased by 3 times, and the incidence has been increasing year by year. It is worth noting that the average age of pancreatic neuroendocrine tumors is only 56.7-13.3 years old, showing a younger trend.

Because most neuroendocrine tumors lack specific manifestations, coupled with unique inert biological characteristics, clinicians often lack understanding, which can easily lead to misdiagnosis and treatment. Taking gastrointestinal pancreatic neuroendocrine tumors (GEP-NEN) as an example, due to the uneven diagnosis and treatment level, GEP-NEN patients may be diagnosed with a delay of up to 7 years. Because of this, as many as 40-95% of GEP-NEN patients have developed distant metastases at the time of diagnosis, and 65-95% of them have liver metastases. Liver metastasis is the most critical prognostic risk factor in GEP-NEN, and it has a decisive impact on the survival of patients. The 5-year survival rate of gastrointestinal neuroendocrine tumors with liver metastasis is 56%-83%, while the 5-year survival rate of pancreatic neuroendocrine tumors is only 48.8%, and the 10-year survival rate is only 30.2%. For limited-stage patients, even if radical surgical resection, up to 94% of cases will still have recurrence and metastasis within 5 years. For inoperable patients, although chemotherapy, targeted therapy, biological therapy and other methods can be used, the effect is still limited. Therefore, the systematic development of basic-clinical translational research on neuroendocrine tumors is very important and imminent.

Based on the above-mentioned problems, this project intends to conduct a systematic and in-depth study of neuroendocrine tumors: 1. Use single-cell sequencing technology to deeply study the molecular biological characteristics of NEN tumors, tumor heterogeneity and cell subtypes. 2. Construct NEN models, including primary cell lines, organoids, and mouse animal models. This study can establish a neuroendocrine tumor research system to find the molecular mechanism and potential intervention targets of NEN recurrence and metastasis, and provide clinicians with safe and effective treatment strategies, thereby improving the therapeutic effect of neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 80, with any gender;
2. Physical fitness score ECOG 0～1 points;
3. The diagnosis is considered as gastrointestinal pancreatic neuroendocrine tumor or pancreatic ductal adenocarcinoma;
4. There is no obvious contraindication to surgery or biopsy;
5. Uncompensated liver cirrhosis, acute and chronic hepatitis and other diseases;
6. No history of other biliary tract related diseases;
7. Volunteer to participate and sign the informed consent form. -

Exclusion Criteria:

1. Patients with non-gastrointestinal pancreatic neuroendocrine tumors or pancreatic ductal adenocarcinoma confirmed pathologically;
2. Suffer from other digestive system diseases, such as irritable bowel syndrome, inflammatory bowel disease;
3. Those who have incomplete follow-up data or refuse to accept follow-up;
4. Patients with other malignant tumors or hematological diseases; -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collect specimens confirmed to be NEN or PDAC by surgery or biopsy histopathology for single-cell sequencing analysis and the construction of primary cells, organoids and animal models.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Bioinformatics analysis of single-cell sequencing results | Half a year
  Analysis of NEN Molecular Biology Information Using Single Cell Sequencing Technology
Model construction | One year
  Collect fresh specimens of NEN to cultivate primary cell lines, construct organoids, and establish animal models of NEN

SECONDARY OUTCOMES:
Exploration of NEN organoid | One year
  To explore and optimize the medium scheme of NEN orgnoid and methods of histomorphological identification of type organs
Tumor microenvironment | One year
  The tumor microenvironment of NEN was analyzed
Comparison of mechanism of NEN with PDAC | Half a year
  Collect fresh specimens of pancreatic ductal adenocarcinoma (PDAC) for single-cell sequencing and organoid construction for comparison with NEN

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Background] Modlin IM, Kidd M, Latich I, Zikusoka MN, Shapiro MD. Current status of gastrointestinal carcinoids. Gastroenterology. 2005 May;128(6):1717-51. doi: 10.1053/j.gastro.2005.03.038. PMID 15887161
- [Background] Dasari A, Shen C, Halperin D, Zhao B, Zhou S, Xu Y, Shih T, Yao JC. Trends in the Incidence, Prevalence, and Survival Outcomes in Patients With Neuroendocrine Tumors in the United States. JAMA Oncol. 2017 Oct 1;3(10):1335-1342. doi: 10.1001/jamaoncol.2017.0589. PMID 28448665
- [Background] Hallet J, Law CH, Cukier M, Saskin R, Liu N, Singh S. Exploring the rising incidence of neuroendocrine tumors: a population-based analysis of epidemiology, metastatic presentation, and outcomes. Cancer. 2015 Feb 15;121(4):589-97. doi: 10.1002/cncr.29099. Epub 2014 Oct 13. PMID 25312765
- [Background] Modlin IM, Oberg K, Chung DC, Jensen RT, de Herder WW, Thakker RV, Caplin M, Delle Fave G, Kaltsas GA, Krenning EP, Moss SF, Nilsson O, Rindi G, Salazar R, Ruszniewski P, Sundin A. Gastroenteropancreatic neuroendocrine tumours. Lancet Oncol. 2008 Jan;9(1):61-72. doi: 10.1016/S1470-2045(07)70410-2. PMID 18177818
- [Background] Saxena A, Chua TC, Sarkar A, Chu F, Liauw W, Zhao J, Morris DL. Progression and survival results after radical hepatic metastasectomy of indolent advanced neuroendocrine neoplasms (NENs) supports an aggressive surgical approach. Surgery. 2011 Feb;149(2):209-20. doi: 10.1016/j.surg.2010.06.008. Epub 2010 Aug 2. PMID 20674950
- [Background] Pape UF, Berndt U, Muller-Nordhorn J, Bohmig M, Roll S, Koch M, Willich SN, Wiedenmann B. Prognostic factors of long-term outcome in gastroenteropancreatic neuroendocrine tumours. Endocr Relat Cancer. 2008 Dec;15(4):1083-97. doi: 10.1677/ERC-08-0017. Epub 2008 Jul 4. PMID 18603570
- [Background] Pavel M, Baudin E, Couvelard A, Krenning E, Oberg K, Steinmuller T, Anlauf M, Wiedenmann B, Salazar R; Barcelona Consensus Conference participants. ENETS Consensus Guidelines for the management of patients with liver and other distant metastases from neuroendocrine neoplasms of foregut, midgut, hindgut, and unknown primary. Neuroendocrinology. 2012;95(2):157-76. doi: 10.1159/000335597. Epub 2012 Feb 15. No abstract available. PMID 22262022
- [Background] Frilling A, Modlin IM, Kidd M, Russell C, Breitenstein S, Salem R, Kwekkeboom D, Lau WY, Klersy C, Vilgrain V, Davidson B, Siegler M, Caplin M, Solcia E, Schilsky R; Working Group on Neuroendocrine Liver Metastases. Recommendations for management of patients with neuroendocrine liver metastases. Lancet Oncol. 2014 Jan;15(1):e8-21. doi: 10.1016/S1470-2045(13)70362-0. PMID 24384494
- [Background] Hanahan D, Coussens LM. Accessories to the crime: functions of cells recruited to the tumor microenvironment. Cancer Cell. 2012 Mar 20;21(3):309-22. doi: 10.1016/j.ccr.2012.02.022. PMID 22439926
- [Background] Baryawno N, Przybylski D, Kowalczyk MS, Kfoury Y, Severe N, Gustafsson K, Kokkaliaris KD, Mercier F, Tabaka M, Hofree M, Dionne D, Papazian A, Lee D, Ashenberg O, Subramanian A, Vaishnav ED, Rozenblatt-Rosen O, Regev A, Scadden DT. A Cellular Taxonomy of the Bone Marrow Stroma in Homeostasis and Leukemia. Cell. 2019 Jun 13;177(7):1915-1932.e16. doi: 10.1016/j.cell.2019.04.040. Epub 2019 May 23. PMID 31130381
- [Background] Ren X, Kang B, Zhang Z. Understanding tumor ecosystems by single-cell sequencing: promises and limitations. Genome Biol. 2018 Dec 3;19(1):211. doi: 10.1186/s13059-018-1593-z. PMID 30509292
- [Background] Heath JR, Ribas A, Mischel PS. Single-cell analysis tools for drug discovery and development. Nat Rev Drug Discov. 2016 Mar;15(3):204-16. doi: 10.1038/nrd.2015.16. Epub 2015 Dec 16. PMID 26669673
- [Background] Lytle NK, Ferguson LP, Rajbhandari N, Gilroy K, Fox RG, Deshpande A, Schurch CM, Hamilton M, Robertson N, Lin W, Noel P, Wartenberg M, Zlobec I, Eichmann M, Galvan JA, Karamitopoulou E, Gilderman T, Esparza LA, Shima Y, Spahn P, French R, Lewis NE, Fisch KM, Sasik R, Rosenthal SB, Kritzik M, Von Hoff D, Han H, Ideker T, Deshpande AJ, Lowy AM, Adams PD, Reya T. A Multiscale Map of the Stem Cell State in Pancreatic Adenocarcinoma. Cell. 2019 Apr 18;177(3):572-586.e22. doi: 10.1016/j.cell.2019.03.010. Epub 2019 Apr 4. PMID 30955884
- [Background] Kumar MP, Du J, Lagoudas G, Jiao Y, Sawyer A, Drummond DC, Lauffenburger DA, Raue A. Analysis of Single-Cell RNA-Seq Identifies Cell-Cell Communication Associated with Tumor Characteristics. Cell Rep. 2018 Nov 6;25(6):1458-1468.e4. doi: 10.1016/j.celrep.2018.10.047. PMID 30404002
- [Background] Sato T, Vries RG, Snippert HJ, van de Wetering M, Barker N, Stange DE, van Es JH, Abo A, Kujala P, Peters PJ, Clevers H. Single Lgr5 stem cells build crypt-villus structures in vitro without a mesenchymal niche. Nature. 2009 May 14;459(7244):262-5. doi: 10.1038/nature07935. Epub 2009 Mar 29. PMID 19329995
- [Background] Jung P, Sato T, Merlos-Suarez A, Barriga FM, Iglesias M, Rossell D, Auer H, Gallardo M, Blasco MA, Sancho E, Clevers H, Batlle E. Isolation and in vitro expansion of human colonic stem cells. Nat Med. 2011 Sep 4;17(10):1225-7. doi: 10.1038/nm.2470. PMID 21892181
- [Background] Karthaus WR, Iaquinta PJ, Drost J, Gracanin A, van Boxtel R, Wongvipat J, Dowling CM, Gao D, Begthel H, Sachs N, Vries RGJ, Cuppen E, Chen Y, Sawyers CL, Clevers HC. Identification of multipotent luminal progenitor cells in human prostate organoid cultures. Cell. 2014 Sep 25;159(1):163-175. doi: 10.1016/j.cell.2014.08.017. Epub 2014 Sep 4. PMID 25201529
- [Background] Chua CW, Shibata M, Lei M, Toivanen R, Barlow LJ, Bergren SK, Badani KK, McKiernan JM, Benson MC, Hibshoosh H, Shen MM. Single luminal epithelial progenitors can generate prostate organoids in culture. Nat Cell Biol. 2014 Oct;16(10):951-61, 1-4. doi: 10.1038/ncb3047. Epub 2014 Sep 21. PMID 25241035
- [Background] Kessler M, Hoffmann K, Brinkmann V, Thieck O, Jackisch S, Toelle B, Berger H, Mollenkopf HJ, Mangler M, Sehouli J, Fotopoulou C, Meyer TF. The Notch and Wnt pathways regulate stemness and differentiation in human fallopian tube organoids. Nat Commun. 2015 Dec 8;6:8989. doi: 10.1038/ncomms9989. PMID 26643275
- [Background] Yoshihara K, Shahmoradgoli M, Martinez E, Vegesna R, Kim H, Torres-Garcia W, Trevino V, Shen H, Laird PW, Levine DA, Carter SL, Getz G, Stemke-Hale K, Mills GB, Verhaak RG. Inferring tumour purity and stromal and immune cell admixture from expression data. Nat Commun. 2013;4:2612. doi: 10.1038/ncomms3612. PMID 24113773